CLINICAL TRIAL: NCT05481398
Title: Negative Pressure Wound Therapy (NPWT) for Incisional Surgical Site Infections in Patients Undergoing Hepatopancreatobiliary Surgery: A Randomized Controlled Trial.
Brief Title: A Randomized Controlled Trial Evaluating the Role of Negative Pressure Wound Therapy (NPWT) for Incisional Surgical Site Infections in Patients Undergoing Hepatopancreatobiliary Surgery
Acronym: NPWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murk Niaz (Other)
Responsible Party: Sponsor-Investigator, Murk Niaz, General Surgery Resident, Sindh Institute of Urology and Transplantation
Organization: Sindh Institute of Urology and Transplantation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NPWT HPB
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Hepatobiliary Disease; Hepatobiliary Disorders; Surgical Site Infection
Keywords: Hepatopancreatobiliary surgery; Surgical site infection; Negative pressure wound therapy
MeSH Terms: conditions — Digestive System Diseases; Surgical Wound Infection | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: Randomization Patients will be randomly allocated into intervention group A (NPWT) or control group (B) by simple randomization.
Who Masked: Outcomes Assessor
Masking Description: Two individuals were assigned the role of outcome assessors to examine the wound after removal of the dressing and score the wound for infection using the ASEPSIS score.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group A (Experimental): After the skin closed, negative pressure wound therapy will be applied.
  Interventions: Other: Negative Pressure Wound Therapy
- Control group B (No Intervention): After the skin is closed, the wound is covered using sterile standard guaze dressing.

INTERVENTIONS:
Other: Negative Pressure Wound Therapy — The wound is dressed using negative pressure wound therapy comprising of a single layer of sterile gauze followed by placement of a 18 Fr nelaton catheter and the wound further covered with 4 more layers of sterile gauze over the nelaton catheter. The wound is then covered with opsite dressing making it airtight. The nelaton catheter is attached to the wall suction port once the patient is shifted to the bed with pressure set at - 25 mm Hg.
  Arms: Intervention group A

SUMMARY:
To compare the rates of incisional surgical site infections (iSSIs) within 7 days of hepatopancreatobiliary (HPB) surgery using negative pressure wound therapy (NWPT) versus using standard sterile gauze dressing.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing elective open HPB surgery (benign or malignant disease) of age > 18 years consenting to the study protocol.

Exclusion Criteria:

The patient in which primary wound closure is not achieved. The patient planned for a second look surgery. The patient with the history of long-term antibiotic use (more than a month). Past history of open abdominal surgery (less than 1 month).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-03-06 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of incisional surgical site infections (iSSIs) | within 7 days of hepatopancreatobiliary (HPB) surgery
  To compare the rates of incisional surgical site infections (iSSIs) within 7 days of hepatopancreatobiliary (HPB) surgery using negative pressure wound therapy (NWPT) versus using standard sterile gauze dressing.

SECONDARY OUTCOMES:
Wound infections | day 7 till 30 days following HPB surgery
  Wound infections after day 7 till 30 days following HPB surgery.
Surgical site complication | within 30 days of HPB surgery
  Surgical site complication (hematoma/seroma/wound dehiscence) within 30 days of HPB surgery.
Rate of fascial dehiscence | within 30 days of HPB surgery
  Rate of fascial dehiscence within 30 days of HPB surgery.
Antibiotic therapy | Day 1 to day 30
  Need for antibiotic therapy for iSSI beyond perioperative/postoperative surgical prophylaxis.
Length of hospital stay. | Day 1 to day 30
  Length of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Uzma Soomro, Principal Investigator — Sindh Institute of Urology and Transplantation
Locations (1):
- Sindh Institute of Urology and Transplantation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided